CLINICAL TRIAL: NCT00618098
Title: A Randomized, Open-label, Efficacy and Safety Study of Octaplex and Fresh Frozen Plasma (FFP) in Patients Under Vitamin K Antagonist Therapy With the Need for Urgent Surgery or Invasive Procedures
Brief Title: Study of Octaplex (Human Prothrombin Complex Concentrate) and Fresh Frozen Plasma in Patients Under Vitamin K Therapy Antagonist Needing Urgent Surgery or Invasive Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEX-205
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Reversal of Anticoagulant Treatment
Keywords: anticoagulant reversal; urgent surgery; invasive procedures; vitamin K; prothrombin complex concentrate
MeSH Terms: conditions — Hemophilia B | interventions — prothrombin complex concentrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Octaplex (human prothrombin complex concentrate) (Experimental): Participants to receive1 or more Octaplex infusions intravenously until their International Normalized Ratio (INR) was < 1.5.
  Interventions: Biological: Octaplex (human prothrombin complex concentrate)
- Fresh frozen plasma (Active Comparator): Participants to receive1 or more fresh frozen plasma infusions intravenously until their International Normalized Ratio (INR) was < 1.5.
  Interventions: Biological: Fresh frozen plasma

INTERVENTIONS:
Biological: Octaplex (human prothrombin complex concentrate) — INR is determined 15 minutes after the end of each infusion. Each dose (mL/kg body weight) was calculated as = ln(INR/1.4)/0.52. The maximum dose for initial treatment was not to exceed 5500 IU. If the INR is ≥ 1.5 after the initial infusion, additional infusions will be repeated until the INR was < 1.5. Octaplex (500 units, IU) is supplied in vials and was reconstituted with 20 mL of Water for Injection (Ph.Eur.).
  Arms: Octaplex (human prothrombin complex concentrate)
Biological: Fresh frozen plasma — INR is determined 15 minutes after the end of each infusion. The initial dose is 10 mL/kg for a participant with an initial INR of < 3 and 15 mL/kg for a participant with an initial INR of ≥ 3. If the INR is ≥ 1.5 after the initial infusion, additional infusions of 5 mL/kg will be repeated until the INR was < 1.5. Fresh frozen plasma is supplied by the blood bank at each study site and will be prepared and handled according to the site's standard practice.
  Other Names: FFP
  Arms: Fresh frozen plasma

SUMMARY:
The purpose of this study is to determine whether Octaplex (human prothrombin complex concentrate) can reverse the effects of anticoagulants when compared to the standard treatment of fresh frozen plasma (FFP).

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate that the efficacy of Octaplex as a reversal agent in patients under vitamin K antagonist therapy with the need for urgent surgery or invasive procedures was not clinically inferior to that of FFP.

The secondary objective of the study is to investigate the safety and tolerability of Octaplex compared to FFP in patients under vitamin K antagonist therapy with the need for urgent surgery or invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age.
* Patients receiving oral anticoagulation with coumadin or warfarin derived agents.
* Patients who have need for urgent surgery or an invasive procedure up to 8 hours after admission or identification of a patient currently hospitalized, where oral or parenteral vitamin K therapy is deemed too slow in its action for reversal of coumadin or warfarin anticoagulant effects.
* Patients with an international normalized ratio (INR) of 2.0 or above.
* Patients who have given written informed consent or for whom written informed consent has been obtained from the patient's legal representative on their behalf.
* Patients able and willing to comply with the procedures laid out in the study protocol. In the case of unconscious and/or incapacitated patients, the willingness of the patient's legal representative for the patient to undergo the procedures laid out in the study protocol.

Exclusion Criteria:

* Patients with a life expectancy of less than 48 hours (eg, patients with a Glasgow Coma Scale (GCS) equal to 3 or a head abbreviated injury score (AIS) of 6, patients requiring continuous inotropic or pressor support, patients status post-cardiac arrest).
* Patients with a history within the last 6 months of disseminated intravascular coagulation (DIC), or hyperfibrinolysis.
* Patients with a known congenital coagulation disorder.
* Patients with known antiphospholipid antibody syndrome or have known lupus anticoagulant antibodies.
* Patients with present or past specific factor inhibitor activity.
* Patients with thrombocytopenia of < 80,000 or a history of heparin induced thrombocytopenia (HIT).
* Patients having received heparin of any type or any non-coumadin or warfarin anticoagulant immediately prior and/or intended to be given within the first 1 hour post-infusion.
* Patients who have received vitamin K more than 3 hours prior to the infusion of study drug.
* Patients with a history of hypersensitivity to plasma-derived products.
* Pregnant or nursing women.
* Patients participating in another clinical treatment study currently or during the past 1 month prior to study inclusion.
* Patients previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, MD, Study Director — International Medical Director
Locations (1):
- Contact Octapharma for Facility details, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octaplex (Human Prothrombin Complex Concentrate) | Fresh Frozen Plasma
Started | 97 | 103
Completed | 66 | 69
Not Completed | 31 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octaplex (Human Prothrombin Complex Concentrate) | Fresh Frozen Plasma | Total
Number analyzed (Participants) | 97 | 103 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.9) | 67.6 (14.8) | 66.6 (19.9)
Age, Customized [Count of Participants; unit: Participants]
  18-60 years | 36 | 30 | 66
  61-74 years | 35 | 34 | 69
  ≥75 years | 26 | 39 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 66 | 71 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian, non-Hispanic | 88 | 96 | 184
  Hispanic | 2 | 3 | 5
  African American | 5 | 4 | 9
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: INR Response
Description: Number of patients who had an INR response, defined as the correction of patient's INR to <1.5, 15 minutes after the end of first infusion with study medication
Time Frame: 15 minutes after the end of first infusion of OCTAPLEX or FFP
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex (Human Prothrombin Complex Concentrate) | Fresh Frozen Plasma
Number analyzed (Participants) | 97 | 103
Participants | 74 | 31

2. Primary Outcome: RBC Transfusion Units
Description: Total number of intra-operative units of red blood cell (RBC) given to patients
Time Frame: Intra-operative; throughout the duration of operation
Measure: Mean (Standard Deviation); unit: mL of RBC Transfusion During Surgery
Groups:
- Octaplex (Human Prothrombin Complex Concentrate)(Pre-interim Analysis): Participants to receive1 or more Octaplex infusions intravenously until their International Normalized Ratio (INR) was < 1.5 and had surgery prior to interim analysis
  Octaplex (human prothrombin complex concentrate): INR is determined 15 minutes after the end of each infusion. Each dose (mL/kg body weight) was calculated as = ln(INR/1.4)/0.52. The maximum dose for initial treatment was not to exceed 5500 IU. If the INR is ≥ 1.5 after the initial infusion, additional infusions will be repeated until the INR was < 1.5. Octaplex (500 units, IU) is supplied in vials and was reconstituted with 20 mL of Water for Injection (Ph.Eur.).
- Fresh Frozen Plasma (Prior to Interim Analysis): Participants to receive1 or more fresh frozen plasma infusions intravenously until their International Normalized Ratio (INR) was < 1.5 and required surgery prior to interim analysis
  Fresh frozen plasma: INR is determined 15 minutes after the end of each infusion. The initial dose is 10 mL/kg for a participant with an initial INR of < 3 and 15 mL/kg for a participant with an initial INR of ≥ 3. If the INR is ≥ 1.5 after the initial infusion, additional infusions of 5 mL/kg will be repeated until the INR was < 1.5. Fresh frozen plasma is supplied by the blood bank at each study site and will be prepared and handled according to the site's standard practice.
- Octaplex (Human Prothrombin Complex Concentrate)(Post-interim Analysis): Participants to receive1 or more Octaplex infusions intravenously until their International Normalized Ratio (INR) was < 1.5 and had surgery post interim analysis
  Octaplex (human prothrombin complex concentrate): INR is determined 15 minutes after the end of each infusion. Each dose (mL/kg body weight) was calculated as = ln(INR/1.4)/0.52. The maximum dose for initial treatment was not to exceed 5500 IU. If the INR is ≥ 1.5 after the initial infusion, additional infusions will be repeated until the INR was < 1.5. Octaplex (500 units, IU) is supplied in vials and was reconstituted with 20 mL of Water for Injection (Ph.Eur.).
- Fresh Frozen Plasma (Post Interim Analysis): Participants to receive1 or more fresh frozen plasma infusions intravenously until their International Normalized Ratio (INR) was < 1.5 and required surgery post interim analysis
  Fresh frozen plasma: INR is determined 15 minutes after the end of each infusion. The initial dose is 10 mL/kg for a participant with an initial INR of < 3 and 15 mL/kg for a participant with an initial INR of ≥ 3. If the INR is ≥ 1.5 after the initial infusion, additional infusions of 5 mL/kg will be repeated until the INR was < 1.5. Fresh frozen plasma is supplied by the blood bank at each study site and will be prepared and handled according to the site's standard practice.
Arm/Group | Octaplex (Human Prothrombin Complex Concentrate)(Pre-interim Analysis) | Fresh Frozen Plasma (Prior to Interim Analysis) | Octaplex (Human Prothrombin Complex Concentrate)(Post-interim Analysis) | Fresh Frozen Plasma (Post Interim Analysis)
Number analyzed (Participants) | 41 | 42 | 56 | 61
mL of RBC Transfusion During Surgery | 0.4 (2.35) | 0.3 (0.77) | 0.2 (0.50) | 0.0 (0.13)

ADVERSE EVENTS:
Time Frame: 21 day Observation Period Post Study Treatment Start (Safety set)
Arm/Group | Octaplex (Human Prothrombin Complex Concentrate) | Fresh Frozen Plasma
All-Cause Mortality (participants affected / at risk) | 19/97 | 13/103
Serious Adverse Events (participants affected / at risk) | 27/97 | 28/103
Other Adverse Events (participants affected / at risk) | 57/97 | 58/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octaplex (Human Prothrombin Complex Concentrate) (N=97) | Fresh Frozen Plasma (N=103)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hemmorhagic Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Failute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Right Ventricular Failure (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Condition Aggravated (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Cardiac Valve Abscess (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis, Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Drug Toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical Device Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Respiratory Distress (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombosis in Device (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Compression (Nervous system disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cardiovascular Insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octaplex (Human Prothrombin Complex Concentrate) (N=97) | Fresh Frozen Plasma (N=103)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 7 (7)
Nausea (Gastrointestinal disorders) | 9 (9) | 13 (13)
Pyrexia (General disorders) | 4 (4) | 7 (7)
Pneumonia (Infections and infestations) | 4 (4) | 7 (7)
Procedural Pain (Injury, poisoning and procedural complications) | 9 (9) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (8) | 6 (6)
Hypotension (Cardiac disorders) | 12 (12) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No